CLINICAL TRIAL: NCT03221387
Title: Feasibility of Using Daily Home HNHF-O2 During Sleep and/or Daytime in Hypercapnic COPD Patients Following Recent (&lt 12 Wks.) Hospitalization for AECOPD for 90 Days
Brief Title: Sleep and Daytime Use of Humidified Nasal High-flow Oxygen in COPD Outpatients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24406
Record Dates: First submitted 2017-07-13; First posted 2017-07-18 (Actual); Results first posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Hypercapnia; Hypoxia
Keywords: Therapy; Noninvasive Ventilation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypercapnia; Hypoxia | interventions — Oxygen Inhalation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Nasal high flow with oxygen (Other): While in the clinic High Flow Nasal Cannula oxygen will be passed through a heated humidifier (AIRVO-2, Fisher and Paykel Healthcare) and applied continuously through large-bore binasal prongs (Optiflow+ Fisher and Paykel Healthcare), with a gas flow rate of 20-35 liters per minute or as high as the patient will tolerate and an FiO2 to keep arterial oxygen saturation (SaO2) > 90%. Temperature will be adjusted based on patient's comfort and range from 34-37 degrees based on prior experience. The subject will be discharged to home and instructed to use the high flow nasal cannula system at night and during the daytime while at home and resting.
  Interventions: Device: Humidified nasal high flow with oxygen

INTERVENTIONS:
Device: Humidified nasal high flow with oxygen — The AIRVO 2 is for the treatment of spontaneously breathing patients who would benefit from receiving high flow warmed and humidified respiratory gases.
  Other Names: AIRVO 2

SUMMARY:
Humidified Nasal High-flow with Oxygen (HNHF-O2) therapy has been reported to have acute beneficial effects in patients with hypoxemic respiratory failure who have been hospitalized. The usefulness of this therapy in the outpatient setting is unproven. This pilot study will test the feasibility of using this therapy in the outpatient setting and its effects on sleep.

DETAILED DESCRIPTION:
Humidified Nasal High-flow with Oxygen (HNHF-O2) therapy has been reported to have acute beneficial effects in patients with hypoxemic respiratory failure. HNHF-O2 may be beneficial in patients with COPD and chronic impairments in gas exchange, both hypoxemia as well as hypercapnia. HNHF-O2 may decrease work of breathing, reduce dyspnea, improve airway humidification, and potentially stabilize or reduce carbon dioxide levels. However, there is limited data showing the chronic effects of HNHF-O2 in patients with hypercapnic respiratory failure, specifically those discharged to home following hospitalization for an acute exacerbation. Data that demonstrates that HNHF-O2 is well tolerated, and stabilizes or improves gas exchange long term in patients with COPD is lacking. Similarly, data that demonstrates that this therapeutic regimen is feasible to provide to patients in the home environment are lacking. This is an open-labeled pilot study of thirty patients to determine the safety and feasibility of using the device in the outpatient management of patients with COPD. A subset of ten patients will have serial sleep studies to determine the effects, if any, on sleep.

ELIGIBILITY:
Inclusion Criteria:

* admitted to the hospital for an acute exacerbation of COPD within the past 12 weeks
* have COPD as the primary diagnosis
* have smoked > 10 pack years.
* receiving supplemental oxygen as part of their usual clinical care.
* willing to give informed consent

Exclusion Criteria:

* upper airway or nasal problems that prohibit the use of high flow oxygen
* current use (≤ 4 weeks of study entry) of any PAP-therapy (e.g., CPAP or NPPV)
* sleep apnea as follows: STOPBang scores ≥ 5 or STOPBang score ≥ 2 plus BMI > 35 kg/m2; or Berlin questionnaire scores suggesting high likelihood of sleep apnea with increased risk of sleep-related accident (e.g., occupation as a commercial driver or pilot);
* excessive daytime sleepiness (i.e., either of High (>15) score on the Epworth Sleepiness Scale or "fall asleep" accident or "near miss" accident in prior 12 months).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-09-10 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard J Criner, MD, Principal Investigator — Temple University Lewis Katz School of Medicine
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nasal High Flow With Oxygen
Started | 30
Completed | 28
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Lung transplant | 1

BASELINE CHARACTERISTICS:
Arm/Group | Nasal High Flow With Oxygen
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] — Self-reported age
  years
    Age | 69.2 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 14
  More than one race | 0
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 14
  More than one race | 0
  Unknown or Not Reported | 1
GOLD grade at enrollment [Number; unit: participants] — GOLD grade is based on FEV1 GOLD 2 Moderate airflow limitation 50% <=FEV1 <80% predicted GOLD 3 Severe airflow limitation 30% <= FEV1 < 50 % predicted GOLD 4 Very severe airflow limitation FEV1 < 30% predicted
  participants
    GOLD 2 | 1
    GOLD 3 | 12
    GOLD 4 | 15

OUTCOME MEASURES:

1. Primary Outcome: Use of Oxygen Therapy by HNHF-O2 at Home
Description: Number of hours of use of the device per day as recorded on the device
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Nasal High Flow With Oxygen
Number analyzed (Participants) | 28
Hours | 6.8 (2.1)

2. Secondary Outcome: Spirometry
Description: Change in FEV1
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Nasal High Flow With Oxygen
Number analyzed (Participants) | 28
Liters | 0.07 (0.6)

3. Secondary Outcome: Change in 6 Minute Walk Distance
Description: Total distance walked in 6 minutes
Time Frame: 90 days
Measure: Mean (Standard Error); unit: meters
Arm/Group | Nasal High Flow With Oxygen
Number analyzed (Participants) | 28
meters | 18.8 (13.6)

4. Secondary Outcome: Breathlessness
Description: Borg dyspnea scale Minimum value =0; Maximum value = 10 Higher scores mean greater shortness of breath
Time Frame: 90 days
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Nasal High Flow With Oxygen
Number analyzed (Participants) | 28
score on a scale | 4.25 (1.1)

5. Other Pre Specified Outcome: Sputum Quantity
Description: Volume of sputum
Time Frame: Measured daily for 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Nasal High Flow With Oxygen
Number analyzed (Participants) | 28
Participants
  No sputum | 15
  1 tbsp or more | 11
  1/4 cup or more | 2

6. Other Pre Specified Outcome: Sputum Consistency
Description: Watery, thin, thick, none, no report made
Time Frame: Measured daily for 90 days
Measure: Number; unit: Daily reports made
Arm/Group | Nasal High Flow With Oxygen
Number analyzed (Participants) | 28
Daily reports made
  None | 838
  Thick | 543
  Thin | 545
  Watery | 182
  No report made | 412

7. Other Pre Specified Outcome: Sputum Color
Description: Clear, yellow, brown, white, none
Time Frame: Measured daily for 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Nasal High Flow With Oxygen
Number analyzed (Participants) | 25
Participants
  None | 12
  White | 8
  Yellow | 3
  Brown | 1
  Green | 1

8. Other Pre Specified Outcome: Peak Flow
Description: liters/minute
Time Frame: Measured daily for 90 days
Measure: Mean (95% Confidence Interval); unit: Liters/minute
Arm/Group | Nasal High Flow With Oxygen
Number analyzed (Participants) | 28
Liters/minute | 243 [239 to 248]

9. Other Pre Specified Outcome: Body Temperature > 100 Degrees F
Description: Yes/no Subjects recorded body temperature via thermometer
Time Frame: Measured daily for 90 days
Measure: Number; unit: percentage of days with fever reported
Arm/Group | Nasal High Flow With Oxygen
Number analyzed (Participants) | 28
percentage of days with fever reported | 15.9

10. Other Pre Specified Outcome: Presence of Cough
Description: Yes/no
Time Frame: Measured daily for 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Nasal High Flow With Oxygen
Number analyzed (Participants) | 28
Participants
  Yes | 9
  No | 19

11. Other Pre Specified Outcome: Presence of Wheeze
Description: Yes/no
Time Frame: Measured daily for 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Nasal High Flow With Oxygen
Number analyzed (Participants) | 28
Participants
  Yes | 13
  No | 15

12. Other Pre Specified Outcome: Presence of Sore Throat
Description: Yes/no
Time Frame: Measured daily for 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Nasal High Flow With Oxygen
Number analyzed (Participants) | 28
Participants
  Yes | 4
  No | 24

13. Other Pre Specified Outcome: Presence of Nasal Congestion
Description: Yes/no
Time Frame: Measured daily for 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Nasal High Flow With Oxygen
Number analyzed (Participants) | 28
Participants
  Yes | 4
  No | 24

14. Other Pre Specified Outcome: Polysomnography
Description: Heart rate
Time Frame: 70 days
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Polysomnography
Description: Pulse oximetry
Time Frame: 70 days
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Polysomnography
Description: Total sleep time in hours
Time Frame: 70 days
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Polysomnography
Description: Sleep efficiency (percent of time sleeping/total amount of time in bed)
Time Frame: 70 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Nasal High Flow With Oxygen
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

LIMITATIONS AND CAVEATS:
Single center study; no active control group; feasibility study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-06): https://cdn.clinicaltrials.gov/large-docs/87/NCT03221387/Prot_SAP_000.pdf